CLINICAL TRIAL: NCT07389317
Title: Assessing the Impact of Illustrated Medication Labels on Medication Understanding Among Migrant and Seasonal Farmworkers in South Georgia
Brief Title: Assessing Illustrated Medication Labels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne Sanderson (Other)
Responsible Party: Sponsor-Investigator, Wayne Sanderson, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 105049; U54OH007547 (NIH)
Record Dates: First submitted 2026-01-23; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Health Behavior; Medication Adherence; Understanding of Medication Instructions
MeSH Terms: conditions — Health Behavior; Medication Adherence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard medication label (Active Comparator)
  Interventions: Behavioral: standard medication label
- Illustrated medication label (Experimental)
  Interventions: Behavioral: Illustrated medication label

INTERVENTIONS:
Behavioral: standard medication label — Standard Education Procedure: Based on best practices, including simple, standardized instructions in the participants' native language and the "teach-back" method.
  Arms: Standard medication label
Behavioral: Illustrated medication label — Illustrated medication labels: Labels will include visuals for medication name, time of administration, food interactions, indications, and potential side effects
  Arms: Illustrated medication label

SUMMARY:
The goal of this clinical trial is to evaluate the impact of graphic-based medication labels on medication understanding and to assess the health literacy of our farmworker population. The main questions it aims to answer are:

Primary Objective: Assess the impact of illustrated medication labels on medication understanding among migrant and seasonal farmworkers Secondary Objective: Evaluate the health literacy of the farmworker population in South Georgia

Participants will be given either medication labels with pictures or standard medication labels

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older
* Receiving medication education at Emory Farm Worker Project (EFP) clinics

Exclusion Criteria:

* Individuals unable to provide informed consent or participate in the study
* Those not requiring medication during their visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2025-05-17 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Medication Understanding Questionnaire (MUQ) | Post intervention (10 minutes)
  MUQ will assess participants' understanding of their medications after education. Scores range from 0-3 to test medication purpose, dose, and frequency

SECONDARY OUTCOMES:
Brief Health Literacy Screen (BHLS) | Post intervention (10 minutes)
  The BHLS consists of 4 questions with each item being worth 1-5 points. Total score range from 4-20 with higher score equating to greater health literacy

CONTACTS AND LOCATIONS:
Overall Officials: Jodie Guest, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University, Atlanta, Georgia
  - University of Kentucky, Lexington, Kentucky

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-09-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT07389317/ICF_000.pdf